CLINICAL TRIAL: NCT06167447
Title: Evaluation Of The Existence Of Kinesiophobia In Patients With Multiple Sclerosis; Effect Of Kinesiophobia On Physical Activity,Functional Status, Quality Of Life and Depression
Brief Title: Evaluation of the Presence and Effects of Kinesiophobia in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Bilge Nur Kilinc, Principal Investigator, Gazi University
Other Study IDs: BNKilinc
Record Dates: First submitted 2023-11-26; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis; Kinesiophobia
Keywords: Multiple sclerosis; kinesiophobia; fear of movement
MeSH Terms: conditions — Multiple Sclerosis; Kinesiophobia | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multiple sclerosis group: Demographic data of all participants were recorded. Tampa Scale of Kinesiophobia (TSK), Beck Depression Inventory (BDI), Quality of Life Scale Short Form-36 (SF-36), International Physical Activity Questionnaire Short Form (IPAQ-SF), Functional Ambulation Classification (FAS), Functional Independence Measure (FIM), Expanded Disability Status Scale (EDSS) were implemented.
  Interventions: Other: questionnaire and examination
- control group: Demographic data of all participants were recorded. Tampa Scale of Kinesiophobia (TSK), Beck Depression Inventory (BDI), Quality of Life Scale Short Form-36 (SF-36), International Physical Activity Questionnaire Short Form (IPAQ-SF), Functional Ambulation Classification (FAS)
  Interventions: Other: questionnaire and examination

INTERVENTIONS:
Other: questionnaire and examination — Demographic data of all participants, height, weight, body mass index, occupation, marriage status, education level, comorbidities, medications used, duration of illness and subtype will be recorded by the researcher. Questionnaires to be filled by patients. On the same day, the musculoskeletal system and neurological examination of the participants will be evaluated by the researcher.

SUMMARY:
The aim of this study was to evaluate the presence of kinesiophobia in multiple sclerosis and to investigate the effect of kinesiophobia on physical activity, functional status, quality of life and depression.

DETAILED DESCRIPTION:
90 people, including 45 patients and 45 healthy control groups, were included in the study. Demographic data of all participants were recorded. Tampa Scale of Kinesiophobia (TSK), Beck Depression Inventory (BDI), Quality of Life Scale Short Form-36 (SF-36), International Physical Activity Questionnaire Short Form (IPAQ-SF), Functional Ambulation Classification (FAS), in addition to Multiple Sclerosis group, Functional Independence Measure (FIM), Expanded Disability Status Scale (EDSS) were implemented.

ELIGIBILITY:
Inclusion Criteria:

* Having a definitive diagnosis of MS according to the 2017 Revised McDonald Diagnostic Criteria
* Expanded Disability Status Scale (EDSS) score between 0-6.5
* Be between the ages of 18-65
* Volunteering to participate in the study

Exclusion Criteria:

* Having orthopedic, psychiatric and other chronic diseases other than MS that may affect physical and cognitive status
* Expanded Disability Status Scale (EDSS) score >6.5
* Being in the MS attack period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 90 people, 45 patients and 45 healthy controls, who applied to the Gazi University Medical School PM&R and Neurology multiple sclerosis outpatient clinic between the ages of 18-65, were included in the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia | through study completion, an average of 6 months.
  Tampa Scale of Kinesiophobia is a checklist of 17 questions developed to measure the fear of movement and re-injury. It is used in many situations such as Acute and chronic pain, Fibromyalgia Syndrome (FMS), musculoskeletal system related injuries, etc. Items in the scale are scored according to a 4-point Likert scoring. A total score of 37 points and above indicates a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Nur Kilinc, Study Director — Gazi University
Locations (1):
- Bilge Nur Kılınç, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dobson R, Giovannoni G. Multiple sclerosis - a review. Eur J Neurol. 2019 Jan;26(1):27-40. doi: 10.1111/ene.13819. Epub 2018 Nov 18. PMID 30300457
- [Background] Zalc B. One hundred and fifty years ago Charcot reported multiple sclerosis as a new neurological disease. Brain. 2018 Dec 1;141(12):3482-3488. doi: 10.1093/brain/awy287. No abstract available. PMID 30462211
- [Background] Walton C, King R, Rechtman L, Kaye W, Leray E, Marrie RA, Robertson N, La Rocca N, Uitdehaag B, van der Mei I, Wallin M, Helme A, Angood Napier C, Rijke N, Baneke P. Rising prevalence of multiple sclerosis worldwide: Insights from the Atlas of MS, third edition. Mult Scler. 2020 Dec;26(14):1816-1821. doi: 10.1177/1352458520970841. Epub 2020 Nov 11. PMID 33174475
- [Background] Kesselring J, Beer S. Symptomatic therapy and neurorehabilitation in multiple sclerosis. Lancet Neurol. 2005 Oct;4(10):643-52. doi: 10.1016/S1474-4422(05)70193-9. PMID 16168933